CLINICAL TRIAL: NCT06723756
Title: A Phase I, Randomized, Double-blind, Single-dose, Partial Replicate, 3-way Cross-over Study to Assess the Total Systemic Exposure Bioequivalence of Budesonide, Glycopyrronium, and Formoterol Delivered by BGF MDI HFO Compared With BGF MDI HFA in Healthy Adult Participants
Brief Title: A Study to Investigate the Exposure of Budesonide, Glycopyrronium, and Formoterol (BGF) Delivered by Hydrofluoroolefin (HFO) Propellant Metered Dose Inhaler (MDI) Compared to a Hydrofluoroalkane (HFA) Propellant MDI in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D598AC00001
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Healthy Participants
Keywords: Asthma; Propellant; Metered dose inhaler
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BGF MDI HFO (Experimental): Participants will receive single doses (2 inhalations as a single dose) of test formulation BGF MDI HFO
  Interventions: Drug: Treatment A: BGF MDI HFO
- BGF MDI HFA (Active Comparator): Participants will receive single doses (2 inhalations as a single dose) of reference formulation BGF MDI HFA
  Interventions: Drug: Treatment B: BGF MDI HFA

INTERVENTIONS:
Drug: Treatment A: BGF MDI HFO — Participants will receive 2 inhalations of BGF MDI HFO (Budesonide/glycopyrronium/fomoterol fumarate pressurized inhalation suspension 160/14.4/4.8 μg per actuation) as a single dose via oral inhalation administered during 1 Treatment period.
  Other Names: Budesonide/glycopyrronium/formoterol fumarate pressurized inhalation suspension, HFO
  Arms: BGF MDI HFO
Drug: Treatment B: BGF MDI HFA — Participants will receive 2 inhalations of BGF MDI HFA (Budesonide/glycopyrronium/fomoterol fumarate pressurized inhalation suspension 160/14.4/4.8 μg per actuation) as a single dose via oral inhalation administered during 2 Treatment periods.
  Other Names: Budesonide/glycopyrronium/formoterol fumarate pressurized inhalation suspension, HFA
  Arms: BGF MDI HFA

SUMMARY:
This study aims to assess the bioequivalence of the total systemic exposure and safety of budesonide, glycopyrronium, and formoterol (160/14.4/4.8 µg/actuation) when administered as BGF MDI HFO compared with BGF MDI HFA in healthy participants.

DETAILED DESCRIPTION:
This is a Phase I, randomized, double-blind, single-dose, single-site, three way cross-over study to assess the pharmacokinetic (PK) and safety of BGF MDI with HFO propellant compared with BGF MDI with HFA propellant in healthy participants (male or female).

The study will comprise of:

* A Screening period of up to 27 days;
* Three Treatment periods: Participants will receive a single dose of the study intervention on three separate occasions (Period 1, Period 2 and Period 3), with the final dose on Day 2 of Treatment Period 3, and a washout period of 5 to 7 days between administration of each dose;
* A final Safety Follow-up within 5 to 7 days after the last administration of the study intervention in Treatment Period 3.

Participants will receive all the treatments as a single dose (2 inhalations) (Treatment A [BGF MDI HFO - test formulation], and Treatment B [BGF MDI HFA - reference formulation]) in one of the 3 possible treatment sequences: ABB, BAB, or BBA. Each participant will be involved in the study for up to 52 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants with suitable veins for cannulation or repeated venipuncture.
* All females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit.
* Females of childbearing potential must not be lactating and if heterosexually active must agree to use an approved method of highly effective contraception.
* Females of non-childbearing potential must be confirmed at the Screening Visit.
* Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 120 kg inclusive.
* Participants must have a forced expiratory volume in the first second (FEV1) ≥ 80% of the predicted normal value (based on age, height, ethnicity and gender at birth) and an FEV1/forced vital capacity (FEV1/FVC) > 70% at the Screening Visit. FEV1/FVC can be reported as ratio ie, 0.7 or a percentage ie, 70%.
* Participants must demonstrate proper inhalation technique and have the ability to properly use an MDI device after training.

Exclusion Criteria:

* History of any clinically significant disease that put the participant at risk of participation.
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, history of narrow angle glaucoma not adequately treated, or bladder neck obstruction/urinary retention.
* Unresectable cancer that has not been in complete remission for at least 5 years.
* Any clinically significant abnormal findings in physical examination, clinical chemistry, hematology, urinalysis results, or vital signs at Screening.
* Any clinically significant abnormalities on 12-lead electrocardiogram (ECG) at Screening.
* Any positive result on Screening for serum hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) antibodies.
* History of any respiratory disorders such as asthma, COPD, or idiopathic pulmonary fibrosis.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity.
* Known or suspected history of alcohol or drug abuse as judged by the Investigator.
* Current smokers or those who have smoked or used nicotine products (including e cigarettes).
* Excessive intake of caffeine-containing drinks or food.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Area under concentration curve from time 0 to the last quantifiable concentration (AUClast) | Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose, and 1, 2, 4, 8, 12 and 24 hours post-dose
Maximum observed drug concentration (Cmax) | Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose, and 1, 2, 4, 8, 12 and 24 hours post-dose

SECONDARY OUTCOMES:
Area under concentration time curve from time 0 to infinity (AUCinf) | Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose, and 1, 2, 4, 8, 12 and 24 hours post-dose
Extrapolated area under the curve from time of last quantifiable concentration (tlast) to infinity, expressed as percentage of AUCinf (AUCextr) | Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose, and 1, 2, 4, 8, 12 and 24 hours post-dose
Time to reach maximum observed concentration (tmax) | Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose, and 1, 2, 4, 8, 12 and 24 hours post-dose
Terminal rate constant (λz) | Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose, and 1, 2, 4, 8, 12 and 24 hours post-dose
Terminal elimination half-life (t1/2λz) | Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose, and 1, 2, 4, 8, 12 and 24 hours post-dose
Mean residence time of the unchanged drug in the systemic circulation from zero to infinity (MRTinf) | Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose, and 1, 2, 4, 8, 12 and 24 hours post-dose
Apparent total body clearance (CL/F) | Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose, and 1, 2, 4, 8, 12 and 24 hours post-dose
Apparent volume of distribution based on the terminal phase (Vz/F) | Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose, and 1, 2, 4, 8, 12 and 24 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: Thank You Card — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D598AC00001&attachmentIdentifier=101207f2-5182-4673-9957-6b35cb8126b3&fileName=2024-10-31_AZ_D598AC00001_TYC_v1.0.pdf&versionIdentifier=